CLINICAL TRIAL: NCT05900102
Title: Evaluating the Current Standard of Care for Patients Diagnosed With Malignant Melanoma of the Head and Neck - Access to Staging and Surgical Treatment
Brief Title: Head and Neck Melanoma; Access to Staging and Surgical Treatment
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Melanoma (Skin); Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Melanoma of the head and neck
- Melanoma of the trunk, arms, or legs

SUMMARY:
Melanoma is a serious type of skin cancer and is the 5th most common cancer in the United Kingdom (UK). It can affect anywhere on the skin including on the head and neck. The cancer often is first noticed as an abnormal mole. Treatment is by removing the cancer with surgery. Early spread of the cancer can be found by testing nearby glands called lymph nodes. This operation is called a sentinel lymph node biopsy (SLNB). If the cancer has spread then new treatments, such as immunotherapy, can be given to help the person live for longer.

The sentinel lymph nodes are usually in the armpits or groin for melanoma on the body, arms or legs. For cancers in the head and neck the sentinel lymph nodes will usually be in the neck. For several reasons SLNB in the neck is not offered in every hospital that manages patients with melanoma. The problem with this is that some patients who could benefit are not offered the new treatments that extend life because it is not known that their cancer has spread.

In this study we aim to gather national data on the management of melanoma of the head and neck including variation in practice between different hospitals. We will use routinely collected anonymous data called 'Hospital Episode Statistics' to look at who is offered SLNB after melanoma of the head or neck, what treatments they have, if their melanoma comes back and how long they survive for.

By doing this, we hope to identify whether SLNB should be made available to everyone diagnosed with melanoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

We will use recorded ICD-10 codes to identify patients for the study. All patients over 18 years of age will be included in the study if they have been coded as:

C43.0 Malignant melanoma of lip C43.1 Malignant melanoma of eyelid, including canthus C43.2 Malignant melanoma of ear and external auricular canal C43.3 Malignant melanoma of other and unspecified parts of face C43.4 Malignant melanoma of scalp and neck C43.5 Malignant melanoma of trunk C43.6 Malignant melanoma of upper limb, including shoulder C43.7 Malignant melanoma of lower limb, including hip

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated by the NHS in England over 18 years of age diagnosed with cutaneous melanoma of the head and neck, and of the trunk or limbs.
Sampling Method: Non-Probability Sample
Enrollment: 86000 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
1. What proportion of patients diagnosed with cutaneous melanoma of the head and neck go on to have SLNB? | 5 years
2. How does this compare to the proportion of patients with cutaneous melanoma in other parts of the body that go on to have SLNB? | 5 years

SECONDARY OUTCOMES:
1. What is the tumour stage of patients with cutaneous melanoma of the head and neck who have SLNB compared to those who do not? | 5 years
2. Do a higher proportion of patients with cutaneous melanoma of the head and neck who have had an SLNB have systemic anti-cancer therapies (or other treatments) for comparable T stage? | 5 years
3. Is there a variation in provision of SLNB for cutaneous melanoma of the head and neck across England? | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Academic Plastic Surgery, Hull University Teaching Hospitals NHS TRust, Cottingham, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No